CLINICAL TRIAL: NCT06922747
Title: FIBROSTEPS Protocol: A 2×2 Factorial Randomized Controlled Trial Evaluating Group Exercise and Somatic Tracking in Fibromyalgia
Brief Title: FIBROmyalgia: Somatic Tracking and Exercise Program Study
Acronym: FIBROSTEPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2025/853403(REK); University of Tromso (Other: University of Tromso)
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Fibromyalgia (FM); Fibromyalgia; Fibromyalgia Syndrome
Keywords: fibromyalgia impact questionnaire; randomized controlled trial; clinical trial; factorial design; 2*2 factorial design; physical activity; somatic tracking; activity; fibromyalgia; pain; effect study; musculoskeletal pain; rheumatic diseases; musculoskeletal diseases
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Pain; Musculoskeletal Pain; Rheumatic Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: The trial applies a 2*2 factorial design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group exercising (Experimental): Receives weekly supervised group exercise sessions, a wrist-worn activity tracker, and access to national recommendations on physical activity.
  Interventions: Other: Group exercising
- Somatic tracking (Experimental): Receives weekly sessions of somatic tracking by a certified therapist, a wrist-worn activity tracker, and access to national recommendations on physical activity.
  Interventions: Other: Somatic tracking
- Group exercising and somatic tracking (Experimental): Receives weekly group exercise sessions, weekly somatic tracking sessions, a wrist-worn activity tracker, and access to national recommendations on physical activity.
  Interventions: Other: Group exercising; Other: Somatic tracking
- Control group (Active Comparator): Receives a wrist-worn activity tracker and access to national recommendations on physical activity.
  Interventions: Other: General activity recommendaitons

INTERVENTIONS:
Other: Group exercising — Weekly, supervised exercise sessions in groups
  Arms: Group exercising; Group exercising and somatic tracking
Other: Somatic tracking — A psychological intervention aiming to learn the brain to reinterpret pain signals.
  Arms: Group exercising and somatic tracking; Somatic tracking
Other: General activity recommendaitons — General recommendaitons for physical activity and healthy lifestyle
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if the combination of two interventions is more effective in treating fibromyalgia symptoms than one intervention alone. The participant group will be people with fibromyalgia in age group 18-65 years. The two interventions to be tested over sixteen weeks are:

* weekly exercise sessions in groups
* weekly consultations with a therapist

The main question it aims to answer is: Is the combination of group exercising and somatic tracking work more efficient than physical activity alone in terms of managing fibromyalgia?

Participants will wear Fitbit activity trackers, register pain intensity daily on a mobile app, and answer the Fibromyalgia Impact Questionnaire (FIQ). They will be divided into four groups:

* one group receiving the exercise intervention
* one group receiving the psychological intervention
* one group receiving both intervention
* one control group recieving general physical activity recommendations

Before the sixteen weeks intervention period, there will be a baseline period of eight weeks. Durng the baseline period, participants will wear activity trackers and maintain their usual lifestyle.

Researchers will compare the combination of the interventions against only one intervention and the control group.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic condition characterised by musculoskeletal pain, fatigue, poor sleep and an overall reduced quality of life. It is well known that physical activity improves symtpons of fibromyalgia, although not all people affected by the condition have positive experiences from exercising. People with fibromyalgia have also stated that physical activity alone is not enough for managing symptomes effectively. This is the background for the proposed randomized controlled trial with a 2*2 factorial design, where two interventions are tested, alone and in combination.

There will be a baseline period of 8 weeks and an intervention period of 16 weeks.

Evaluations will occur at the end of the baseline period (8 weeks) and at the end of the intervention period (24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with fibromyalgia according to the criteria specified in Wolfe et al (2016)
* Able to perform light physical activity
* Able to provide written informed consent
* Owning a smartphone
* Able to be followed for 24 weeks

Exclusion Criteria:

* Pregnant
* Severe co-morbid psychiatric or neurological disorders
* Current participation in another clinical trial
* Recent surgery or other physical constraints preventing exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Total FIQ score | At end of baseline (8 weeks) and post-intervention (24 weeks)
  Fibromyalgia Impact Questionnaire (FIQ) is widely used in clinical trials in fibromyalgia patients. The questionnaire contains questions that are answered using a scale. The scores from each question are used to calculate a total FIQ score.

SECONDARY OUTCOMES:
Steps per day | 24 weeks
  Measured by Fitbit activity trackers
Resting heart rate | 24 weeks
  Measured by Fitbit
Insomnia Severity Index (ISI) | At end of baseline (8 weeks) and post-intervention (24 weeks)
  ISI is calculated from a questionnaire containing sleep and insomnia related questions
Self-reported pain intensity | 24 weeks
  Self-reported pain intensity measured by Visual Analogue Scale (VAS). Participants will be asked to register their pain intensity once daily through a mobile application.
Minutes lightly active | 24 weeks
  Measured by Fitbit
Minutes moderately active | 24 weeks
  Measured by Fitbit
Minutes very active | 24 weeks
  Measured by Fitbit
Sleep efficiency | 24 weeks
  Measured by Fitbit. The formula for sleep efficiency is time asleep/(total time in bed - time to fall asleep)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tromsø, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No